CLINICAL TRIAL: NCT06136130
Title: The Effect of Positioning With Material and Hand-Face Maneuver on Physiological Parameters and Stress Symptoms in Preterm Newborns
Brief Title: The Effect of Positioning With Material and Hand-Face Maneuver
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran University (Unknown)
Responsible Party: Principal Investigator, Isıl AR, Research Assistant, Kirsehir Ahi Evran University
Organization: Kirsehir (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IAR
Record Dates: First submitted 2022-12-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Stress; Position
Keywords: preterm; position; stress; physiological parameters
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The Effect of Positioning with Material and Hand-Face Maneuver on Physiological Parameters and Stress Symptoms in Preterm Newborns
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positioning Material (Experimental): Preterm infants in Intervention group were placed in the nest with positioning material and placed in lateral and prone positions
  The positioning material and hand-face maneuver were applied together to the preterm infants in the intervention group, and they were given lateral and prone positions in this way in the second day
  Interventions: Device: Tortoise Positioning Material Group
- Standard Care (No Intervention): Standard care was used

INTERVENTIONS:
Device: Tortoise Positioning Material Group — Preterm infants were placed in the nest with positioning material and placed in lateral and prone positions The positioning material and hand-face maneuver were applied together to the preterm infants in the Positioning Material Group 2, and they were given lateral and prone positions in this way
  Other Names: Control Group
  Arms: Positioning Material

SUMMARY:
The study was administered in a randomized controlled experimental design to evaluate the effects of material positioning and hand-face maneuver on physiological parameters and stress symptoms in preterm newborns with gestational weeks 28 to 32. The sample of the study consisted of 60 preterm infants who met the selection criteria in newborn intensive care unit between September 2018 and July 2020.The newborns in the control group (n=30) were given a "nesting with a rolled up blanket" position, as in the routine of the ward. The Experimental Group1 (n=30) was given positions using a "positioner" and the same newborns (Experimental2) was given positions using "positioner and hand-face maneuver" on the second day of the study.

DETAILED DESCRIPTION:
The universe of the study consisted of preterm newborns patients who met the selection criteria in newborn intensive care unit.The research was planned as a randomized controlled experimental study. In order for the groups to be distributed homogeneously, the order produced by a computer program (http://www.randomizer.org/) was used. Patients who meet the inclusion criteria and agree to participate in the study assigned to the experimental and control groups according the randomization list. The control variable of the study is demographic characteristics of the baby. The dependent variables of the study are physiological parameters, newborn position assesment tool score and newborn stress scale score In the research, "Information and follow-up form" prepared by the researcher in line with the literature was used as data collection tools. Newborn Position Assesment Tool and Newborn Stress Scale were also used

ELIGIBILITY:
Inclusion Criteria:

* Preterm newborn between 28-32 weeks of gestation (very early preterm)
* Not connected to mechanical ventilator
* Parent's consent with informed consent form

Exclusion Criteria:

* Presence of congenital anomalies, a known infection, neuromuscular problems and genetic anomalies in a preterm newborn
* Have undergone any surgical intervention
* Painful procedure (invasive procedure, etc.) performed in the last hour
* Taking analgesics in the last six hours

Ages: 28 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Newborn Position Assesment Tool | Before starting position, after 1 hour 1st position , before second positon, after 1 hour second position
  The Infant Position AssessmentTool (IPAT) is a six-item(shoulders, hands, hips, knees,ankles, feet, head, neck) tool with cumulative scores ranging from 0 to 12. A scale score of 12 indicates that the position is given very well, and a score of 0 indicates that the position is very bad.
Newborn Stress Scale | Before starting position, after 1 hour 1st position , before second positon, after 1 hour second position
  Scale items were collected in 8 subgroups. These subgroups consist of a total of 24 items in 3-point Likert type, including facial expression, body color, respiration, activity level, comfortability, muscle tone, extremities, and posture.A minimum of 0 points and a maximum of 16 points are taken from the scale. As the score increases, the baby's stress level increases.
Pulse rate assesment | Before starting position, after 1 hour 1st position , before second positon, after 1 hour second position
  Pulse rate/min
Respiratory rate assesment | Before starting position, after 1 hour 1st position , before second positon, after 1 hour second position
  respiratory rate/min,
Oxygen saturation assesment | Before starting position, after 1 hour 1st position , before second positon, after 1 hour second position
  Oxygen saturation %

CONTACTS AND LOCATIONS:
Overall Officials: Serap Balcı, Assoc. Prof., Study Director — İstanbul University Cerrahpaşa; Isil AR, PhD, Study Chair — İstanbul University Cerrahpaşa
Locations (1):
- Kocaeli University Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ar I, Balci S. The effect of the use of positioning materials and hand-face maneuvers on physiologic parameters and stress symptoms in preterm newborns. Ital J Pediatr. 2025 Jul 21;51(1):239. doi: 10.1186/s13052-025-02070-z. PMID 40691617